CLINICAL TRIAL: NCT05703022
Title: Early Exercise Training in Patients Following Heart Valve Surgery for Infective Endocarditis. A Feasibility Study.
Brief Title: Early Exercise Training in Patients Following Heart Valve Surgery for Infective Endocarditis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: UiT The Arctic University of Norway (Other); Herlev and Gentofte Hospital (Other); Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Interventional
Record Dates: First submitted 2021-10-12; First posted 2023-01-27 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Endocarditis; Heart Valve Diseases
Keywords: Training; Heart valve surgery; Infective endocarditic
MeSH Terms: conditions — Endocarditis; Heart Valve Diseases

STUDY DESIGN:
Intervention Model Description: Single centre feasibility study to assess acceptability, compliance, delivery of the intervention and expected effect sizes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early exercise training (Experimental): Supervised aerobic interval training (uphill treadmill walking or cycling on an exercise bike 4x4 min at 65-85% of peak heart rate) 3 times weekly.
  Interventions: Other: Aerobic interval training

INTERVENTIONS:
Other: Aerobic interval training — The intervention will start between 7 and 21 days after heart valve surgery. While hospitalized the participants will perform supervised aerobic interval training comprised 4x4 minute, 3 times per week. Intensity will start at 60% of maximum heart rate in the first week, around 13-14 in Borg RPE-Scale. The workload will be gradually increased as the participant tolerance improves, but not above 85% of maximum heart rate or 16-17 in Borg RPE Scale.

SUMMARY:
A prospective, interventional, single-group, single centre study to evaluate the feasibility of early aerobic exercise training in patients following heart valve surgery for infective endocarditis.

DETAILED DESCRIPTION:
Infective endocarditis (IE)is uncommon, but people with some heart conditions have a greater risk of developing it. Well designed studies have shown that the majority of the IE population have low physical function and many are inactive. This is negative for their health and well-being. High-intensity aerobic interval training has shown to be beneficial in patients with other cardiovascular disorders. Presumably, patients with IE also benefit from such treatment, but the optimal training mode,intensity, frequency and duration to improve aerobic capacity are not clear. This study will explore how aerobic interval training supported by smartwatch may contribute to the physical activity after infective endocarditis . Throughout the project, investigators will explore opportunities and barriers for supervised individualised exercise training for IE patients that has been treated with heart valve surgery.

The primary objective is to explore how early aerobic interval training can be safely performed and accepted in patients with infective endocarditis after heart valve surgery. The two main research questions are:

1. How is aerobic interval training experienced by patients with IE after heart-valve surgery?
2. Can aerobic interval training with smartwatch support be accepted and safely performed by patients who have undergone endocarditis and left-sided heart-valve surgery?

The study is a single centre feasibility study, at the University Hospital of North Norway in Tromsø .The study duration from the first assessment of the first patient to the last assesment of the last patient: 24 months. The in-hospital training intervention for each patient will start between 7 and 21 days after the heart valve surgery and continue in university or local hospital for 3 months.

Investigators will recruit between 10 and 20 participants from the University Hospital of North Norway.

ELIGIBILITY:
Inclusion Criteria:

* (1)patients presenting with confirmed infectious endocarditis, with left-sided heart valve surgery and without arterial embolus,
* (2)being residents of Northern Norway,
* (3)willing and able to give informed consent 4-21 days after the heart valve surgery.

Exclusion Criteria:

* (1)patients who are hemodynamically or respiratory unstable, have temperature > 38 or positive blood cultures
* (2)clinically significant serious concurrents medical condition such as premorbid illnesses and other concurrens serious infection which could affect the safety or tolerability of the intervention
* (3)clinically significant concurrens musculoskeletal disorder or other concurrent disease or injury that may inhibit physical activity.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Feasibility of inhospital aerobic interval training | 3 months
  Number of completely finished training sessions will be record.
Experience with inhospital aerobic inetrval training assessed by semi structured interviews | Before discharge
  Semi structured interviews will involve patients opinions on the strengths and weaknesses of the inhospital training intervention.
Experience with inhospital aerobic inetrval training assessed by semi structured interviews | 3 months
  Semi structured interviews will involve patients experiences of adopting and following the trainings program at home.

SECONDARY OUTCOMES:
Intervention related endpoints 1 | During intervention
  Number of training sessions
Intervention related endpoints 2 | During intervention
  Duration of training sessions
Intervention related endpoints 3 | During intervention
  Intensity of training sessions: Speed on the treadmill, bicycel or step box
Intervention related endpoints 4 | During intervention
  Exercise method.
Patient related endpoints 1 | During intervention
  Peak heart rate measured with Apple Watch
Patient related endpoints 2 | During intervention
  Atrial fibrillation episodes will be measured with Apple Watch
Patient related endpoints 3 | During intervention
  Blood pressure wil be measured before and after training sessions
Patient related endpoints 4 | During intervention
  Borg RPE-Scale
Sub-maximal oxygen uptake | Sub-maximal oxygen uptake at 2 weeks
  A graded treadmill test of sub-maximal oxygen uptake using a breath by breath ergospirometer
Sub-maximal oxygen uptake | Sub-maximal oxygen uptake at 3 months
  A graded treadmill test of sub-maximal oxygen uptake using a breath by breath ergospirometer
6 minute walk test | 6 minute walk test at 2 weeks
  Walking distance (in meters) will be measured with the 6 minute walk test
6 minute walk test | 6 minute walk test at 3 months
  Walking distance (in meters) will be measured with the 6 minute walk test
Physical Activity | Physical activity 2 weeks
  Axivity AX3 Accelerometers
Physical Activity | Physical activity 3 months.
  Axivity AX3 Accelerometers
Experience with inhospital aerobic - Questionaire | Before discharge
  The questionnaire will contain validated questions from the PasOpp questionnaire along with questions specifically prepared for this study on process and experience outcomes.
Experience with inhospital aerobic - Questionaire | 3 months.
  The questionnaire will contain validated questions from the PasOpp questionnaire along with questions specifically prepared for this study on process and experience outcomes.
Physical Activity | Physical activity at 2 weeks
  Apple Watch
Physical Activity | Physical activity at 3 months
  Apple Watch

OTHER OUTCOMES:
HeartQOL | Changes from baseline in heart /health-related quality of life at 3 months
  Health-related quality of life assessed by The Norwegian version of Heart QOl for patients with coronary heart disease with scale 0-3, where 3= A lot heart problems and 0=No problems
EQ5D-5L | Changes from baseline in health-related quality of life at 3 months
  Health status assessed by The Norwegian version of EQ-5D-5L with EQ Visual Analogue scale (EQ VAS) 0-100, where 0=worst health and 100=best health
New cardiovascular or cerebrovascular incidents. | 3 months
  Gathered from participants and their electronic journal system

CONTACTS AND LOCATIONS:
Overall Officials: Gyrd Thrane, PhD, Study Chair — UiT The Arctic University of Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No